CLINICAL TRIAL: NCT00449124
Title: A Phase I, Randomized, Double-Blind, Dose-Ranging, Crossover Trial of HCV Vaccine (TG4040) in Patients With Chronic Hepatitis C to be Conducted in Two Parts
Brief Title: TG4040 in Patients With Chronic HCV
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 05-0061
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2008-06

CONDITIONS: Hepatitis C
Keywords: hepatitis C, vaccine, TG4040
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Part I-group 1 (Experimental): Part I/Group 1: Cycle 1-TG4040 10^6 PFU days 0, 7 and 14; Cycle 2-Placebo days 0, 7 and 14; Cycle 3-Placebo days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040
- Part IIa-group 1 (Experimental): Part IIa/Group 1: Cycle 1-TG4040 10^8 PFU days 0, 7 and 14; Cycle 2-Placebo days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040
- Part IIa-group 2 (Experimental): Part IIa/Group 2: Cycle 1-Placebo days 0, 7 and 14; Cycle 2-TG4040 10^8 PFU days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040
- Part I-group 3 (Experimental): Part I/Group 3: Cycle 1-Placebo days 0, 7 and 14; Cycle 2-Placebo days 0, 7 and 14; Cycle 3-TG4040 10^8 PFU days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040
- Part I-group 2 (Experimental): Part I/Group 2: Cycle 1-Placebo days 0, 7 and 14; Cycle 2-TG4040 10^7 PFU days 0, 7 and 14; Cycle 3-Placebo days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040
- Part IIb-group 1 (Experimental): Part IIb/Group 1: Cycle 1-TG4040 10^8 PFU days 0, 7 and 14; Cycle 2-Placebo days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040
- Part IIb-group 2 (Experimental): Part IIa/Group 2: Cycle 1-Placebo days 0, 7 and 14; Cycle 2-TG4040 10^8 PFU days 0, 7 and 14.
  Interventions: Drug: Placebo; Biological: TG4040

INTERVENTIONS:
Drug: Placebo — Injections of 0.5 mL of normal saline solution (0.9% NaCl).
Biological: TG4040 — Modified vaccinia virus Ankara encoding hepatitis C virus (HCV) proteins NS3, NS4, and NS5B administered by subcutaneous injection into the thigh. Dosages: TG4040 10^6 PFU, TG4040 10^7 PFU and TG4040 10^8 PFU.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an investigational vaccine (TG4040) to prevent hepatitis C virus (HCV) infection. The primary goal of this study is to determine the safety of increasing doses of TG4040 versus placebo (an inactive substance) in subjects chronically infected with HCV. Approximately 85 patients, ages 18-65 years, with chronic HCV infection will be enrolled in this study at two sites, Saint Louis University and Cincinnati Children's Hospital. Volunteers will receive doses of TG4040 and placebo by injections into the thigh on different days, depending on which study group they belong to. Safety will be checked before doses are increased, and each participant will receive the study vaccine, TG4040, at some point during the study. Each subject will participate in the study for 8 months. This study may help produce a new vaccine that would improve control of HCV.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, immunogenicity, and efficacy of the hepatitis C virus (HCV) vaccine, TG4040, in outpatients with chronic hepatitis C. The study will be conducted in two parts at two DMID Vaccine Treatment and Evaluation Unit (VTEU) Centers: Saint Louis University and Cincinnati Children's Hospital. Up to 85 subjects with chronic hepatitis C will receive the test vaccine via subcutaneous injection into the thigh. In Part I of this study, 18 subjects will be randomized to 1 of 3 groups. At the initial dosing time point, Group One will receive 10 to the 6th power particle-forming units (PFU) and Groups Two & Three will receive saline placebo in 3 doses on Days 0, 7, and 14. After Safety Monitoring Committee (SMC) review, Group Two will receive a higher dose of TG4040 (10 to the 7th power PFU) and Groups One & Three will receive saline placebo. After a further SMC review, Group Three will receive a higher dose of TG4040 (10 to the 8th power PFU) and Groups One & Two will receive saline placebo. (Each subject will therefore be treated with one course of TG4040 and receive two courses of placebo). In Part II of this study, 60 subjects (30 non-responders or relapse subjects-Part IIa, and 30 treatment naïve, Part IIb) will be randomized into two groups to receive either 10 to the 8th power PFU (or the highest tolerated dose) of TG4040 or saline placebo at two dosing time points with a crossover design. (Each subject will therefore be vaccinated with the same dose of TG4040 and also receive a course of placebo.) Subjects enrolled in either Part I or Part II of the study will participate for 8 months. The primary objective for Part I of the study is to assess the safety of escalating doses of TG4040 versus placebo administered to non-responders or relapse subjects with chronic hepatitis C. The secondary objective for Part I of the study is to assess immunogenicity of escalating doses of TG4040 versus placebo administered to non-responders or relapse subjects with chronic hepatitis C. The primary safety objective for Part II of the study is to assess the safety of the dose of TG4040 selected from Part I versus placebo when administered to subjects with chronic hepatitis C, either non-responders or relapse subjects or treatment- naïve subjects. The primary efficacy objective for Part II of the study is to assess antiviral activity against HCV of TG4040 versus placebo in subjects with chronic hepatitis C, non-responders or relapse subjects or treatment-naïve subjects, assessed as a 1 log reduction in serum level of HCV RNA. The secondary objective for Part II of the study is to assess immunogenicity of TG4040 versus placebo in subjects with chronic hepatitis C, non-responders or relapse subjects or treatment-naïve subjects, and correlate this with reductions in serum levels of HCV RNA. For Part I, the primary outcome measures are related to safety and include measures of reactogenicity, changes in blood counts and hepatic panel. For Part II, the primary outcome variable is a change in serum levels of HCV RNA compared to baseline. A decrease in more than 1 log from baseline will be considered a significant effect. In addition to this, other primary outcome measures will also include safety and include measures of reactogenicity, changes in blood counts and hepatic panel. Secondary outcomes measures include those tests aimed at assessing immunogenicity of the vaccine candidate and include, but are not limited to, development of anti-HCV using standard commercial assays and research assays, developed of enhanced in vitro T cell reactivity when stimulated with HCV antigens.

ELIGIBILITY:
Inclusion Criteria:

Part I and Part II:

1. Informed consent obtained and signed;
2. Male or female patients, age 18-65 years old (inclusive)
3. Female patients will be menopausal for at least 12 months, surgically sterile or agree not to become pregnant from the time of study enrollment until at least 28 days after the administration of vaccine or placebo. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized.

   If the volunteer is female, of childbearing potential, and sexually active, she agrees to use acceptable contraception. (Acceptable contraception methods are restricted to effective intrauterine devices (IUDs) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination and for the entire study period post-vaccination).

   Note: A woman is eligible if she is monogamous with a vasectomized male or abstinent, without the additional need for hormonal or barrier birth control methods upon review of a reproductive history.
4. With chronic hepatitis C evidenced by:

   * HCV RNA detectable in blood, and
   * A liver biopsy compatible with chronic hepatitis C;
5. Infected with HCV genotype 1;
6. Non-cirrhotic patients, i.e. liver biopsy available within one year prior to baseline, excluding stage 4 fibrosis; otherwise, if no liver biopsy of less than one year is available, it will be performed at baseline;
7. Patients participating in:

   * Part I will be non-responder patients: patients having received at least 3 months of pegylated IFN-alpha (IFN-alpha) plus ribavirin, with currently detectable HCV RNA (whether or not they reach, Early Virologic Response (EVR, defined as a reduction of HCV RNA by at least 2 logs from baseline or negative at 12 weeks) and/or SVR) with > 6 months between the end of PEG IFN-alpha treatment and the first TG4040 injection;
   * Part IIa will be either non-responder or relapser patients. Part IIb will be treatment-naïve patients: patients who have never received IFN-based treatment
8. Patients must have compensated liver disease, defined through use of the Child-Pugh scoring system with:

   * Features of low serum albumin, prolonged prothrombin time, raised bilirubin, ascites and hepatic encephalopathy are scored and patients assigned to Child-Pugh class A, B or C, the later two being decompensated. Only patients with compensated liver disease will be enrolled.
   * No history of ascites, hepatic encephalopathy or bleeding from esophageal varices laboratory tests values:
   * Serum bilirubin and international normalized ratio (INR) values <1.2 (except in patients with Gilbert syndrome where serum bilirubin may be as high as 3.0 mg/dL)
   * Serum alanine aminotransferase (ALT) < 5 fold the upper limits of normal (ULN) and
   * Other laboratory parameters of grade 0 or 1 (CTC criteria)

Exclusion Criteria:

Part I and Part II:

1. Co-infection with HBV (indicated by the presence of hepatitis B surface antigen (HBsAg) in serum) or HIV (anti-HIV in serum); patients with HIV positive sexual partner (by history) will not be included;
2. Current HCV therapies through out the trial period
3. Current alcohol abuse or drug addiction that in the opinion of the investigator may interfere with the subject's ability to comply with trial procedures.
4. History of immunodeficiency
5. Known or suspected impairment of immunologic function including moderate to severe kidney impairment
6. Malignancy within the last 5 years, not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site
7. Significant cardiac disease, evidenced by:

   * History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, chest pain or shortness of breath on activity, or other heart conditions under the care of a physician
   * Baseline ECG showing clinically significant abnormalities (e.g., all kinds of advanced atrioventricular block or intraventricular block with QRS >120msec, QTc >460 msec, or frequent premature atrial contractions, atrial fibrillation or other atrial arrhythmias, > ventricular couplets or ST-T wave abnormalities diagnostic of myocardial ischemia or prior myocardial infarction. EKGs will be interpreted by an identified cardiologist at Saint Louis University prior to enrollment.
   * Baseline echocardiogram showing clinically significant abnormalities including valvular disease or contractile dysfunction.
   * Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp)

   NOTE: This criterion applies only to subjects 20 years of age and older AND only if at least one of the following apply:

   A) have smoked a cigarette in the past month, and/or B) have hypertension (defined as systolic blood pressure >140 mm Hg) or are on antihypertensive medication, and/or C) have a family history of coronary heart disease in male first-degree relative (father or brother) < 55 years of age or a female first-degree relative (mother or sister) < 65 years of age.
8. Current use of immunosuppressive medication; Corticosteroid nasal sprays, Inhaled steroids for asthma and/or topical steroids are permissible. Persons taking short courses of oral steroids for conditions such as poison ivy will need to wait a period of 2 weeks after completion of the steroids to begin vaccination.
9. History of any one of the following:

   * Suicide attempt or hospitalization for depression within the past five years.
   * Any current (within 6 months) severe or poorly-controlled psychiatric disorder (e.g., depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, personality disorder).
   * The following patients must be excluded unless they are assessed and followed by a psychiatrist or other mental health professional who pre-approves their study participation:
   * Patients who have had a suicide attempt and/or hospitalization for depression more than 5 years ago.
   * Patients who have had a severe or poorly-controlled psychiatric disorder (e.g., depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, personality disorder) more than 6 months ago but less than 5 years ago.
10. Receipt of any inactivated vaccine 14 days prior to vaccination or for the duration of the study
11. Receipt of any live attenuated vaccine within 30 days prior to vaccination or for the duration of the study
12. Receipt of any MVA vaccine in the last five years
13. Use of any experimental agent within 30 days prior to vaccination or for the duration of the study
14. Receipt of blood products or immunoglobulin within six months prior to vaccination
15. Donation of a unit of blood within 56 days prior to vaccination or for the duration of the study following the first vaccination
16. Acute febrile illness (>100.5 degrees F) on the day of vaccination
17. Pregnant or lactating women
18. Any condition that, in the opinion of the investigator, might interfere with study objectives
19. Known allergy to MVA vaccine
20. Receipt of antiviral drugs such as alpha interferon or ribavirin
21. Other laboratory parameters of grade 2 or more
22. Study personnel engaged in the blinding of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2007-09 (Estimated); Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Part I and Part II: safety including measures of reactogenicity, changes in blood counts and hepatic panel. | Solicited reactogenicity and AEs will be collected on the day of vaccination and daily for 6 days following vaccination. Unsolicited AEs will be collected throughout the study period.
Part II: change in serum levels of HCV RNA compared to baseline. | Part I: screening days -60 and -30, days 0, 14, 28 and month 6. Part II: screening days -60 and -30, days 0, 14, 28, 56, 90, and 180.

SECONDARY OUTCOMES:
Tests to assess immunogenicity of the vaccine candidate and include, but are not limited to, development of anti-HCV using standard commercial assays and research assays, developed of enhanced in vitro T cell reactivity when stimulated with HCV antigens. | Part I: time points 1, 2, and 3-days 0, 7 and 14 post-vaccination and 2 months following the 3rd vaccination. Part II: time points 1 and 2-days 0, 7 and 14 post vaccination and 1, 2, 3 and 6 months following the 2nd vaccination.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio